CLINICAL TRIAL: NCT05220696
Title: Central Venous Oxygen Saturation and Carbone Dioxide (CO2)-Derived Indices in the Critically: Correlation of Measurements According to the Site of Harvest (Femoral Versus Jugular Vein)
Brief Title: Central Venous Oxygen Saturation and Carbone Dioxide (CO2)-Derived Indices in the Critically:
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL22_0003
Record Dates: First submitted 2022-01-17; First posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Shock
Keywords: Adult > 18 YO; Venous catheter in femoral and jugular sites; Arterial catheter; central venous to arterial carbon dioxide difference; central venous to arterial carbon dioxide difference to arterial to venous oxygen difference; central venous oxygen saturation
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — NC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill patients with shock: Critically ill patients with shock

SUMMARY:
The optimal management of shock states requires a precise evaluation of several parameters, clinical, biological, hemodynamic, and echocardiographic. Among these, parameters that measure O2 and CO2 consumption are of a great interest, especially PCO2 arteriovenous gradient (PCO2 gap) and O2 arteriovenous difference [D(a-v) O2]. The PCO2 gap best correlates with cardiac output while the PCO2gap/D(a-v)O2 ratio would be earlier and more specific than blood lactate assay in assessing tissue hypoperfusion secondary to shock.

The PCO2 gap and the PCO2gap/D (a-v) O2 ratio have been evaluated from gas measurements of venous blood collected from the pulmonary artery and from the superior vena cava area. However, in some patients the placement of a catheter in the superior vena cava is difficult or even impossible due to thrombosis, vascular occlusions and other reasons… In these cases, the inferior vena cava is used for drugs infusion, nutrition and possibly samples. Gasometric samples in lower cellar territory have not yet been validated and may not be correlated with measurements in upper cellar territory. It is therefore useful for current practice to validate samples in lower cellar territory and demonstrate their correlation with measurements made in upper cellar territory.

During an observation period, in patients with catheters in the superior and inferior vena cava for therapeutic indications (renal replacement therapy,...), the investigators systematically took gas measurements at the femoral and jugular sites. the investigators used these data to assess the correlation of PCO2 gap measurements and carbon dioxide-derived indices according to the harvest site : jugular and femoral venous.

ELIGIBILITY:
Inclusion criteria:

- All consecutive critically ill patients who had an arterial catheter and a venous catheter in the superior and inferior vena cava were included.

Exclusion criteria:

* An age under 18
* Pregnancy
* Legally protected adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
The correlation of the measurement of indices derived from carbon dioxide (CO2) | day 1
  To assess the correlation of the measurement of indices derived from carbon dioxide (CO2) according to the femoral or jugular harvest site in the critically ill patient. Measurements included venous pCO2 and pO2, and central venous saturation ; arterial pO2 and pCO2.
  From these measurements, carbon dioxides and oxygen variables were calculated as follows :
  PCO2gap= Pv-aCO2= PvCO2 -PaCO2, where PaCO2 and PvCO2 represent their arterial and venous partial pressures respectively D(a-v)O2= CaO2- CvO2= [(hg x SaO2 x 1.34) + (Pa02 x O.OO3)]- [(hg x SvO2 x 1.34) + (Pv02 x O.OO3)], where CaO2 and CvO2 are the arterial and venous 02 content, PaO2 and PvO2 represent their arterial and venous partial pressures respectively.
  Venous measurements are realized in both venous jugular and femoral sites.

SECONDARY OUTCOMES:
To assess the correlation of the measurement of venous O2 saturation | day 1
  To assess the correlation of the measurement of venous O2 saturation according to the femoral or jugular harvest site. To find a simple equation allowing to calculate the gasometric parameters superior vena cava PCO2 gap and ratio PCO2gap / D (a-v) O2 from measurements made at the femoral level

CONTACTS AND LOCATIONS:
Overall Officials: Kada KLOUCHE, MD PhD, Study Director — UH Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC